CLINICAL TRIAL: NCT06900699
Title: Clinico-pathological Features and Outcomes of High Risk Gestational Trophoblastic Neoplasia Patients: an Observational Cross-sectional Study
Brief Title: Clinicopathological Features , Outcomes and Prognostic Factors of High Risk Patients of Gestational Trophoblastic Neoplasia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Neveen Adel Aness Zakhari, resident, Assiut University
Other Study IDs: GTN high risk patient
Record Dates: First submitted 2025-03-16; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Gestational Trophoblastic Neoplasias (GTN)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- high risk GTN patients according WHO classification: there is no interventions

SUMMARY:
Aim of the Study This study aims to investigate the clinical and pathological features, treatment outcomes, and prognostic factors in high-risk patients with Gestational Trophoblastic Neoplasia (GTN).

Objectives:

* Identify common clinical and pathological features of high-risk GTN patients.
* Required surgical treatment as primary or subsequent line.
* Evaluate how well different treatments work and their side effects.
* Find factors that can help predict patient outcomes.
* Compare survival rates and relapse risks among patients.

DETAILED DESCRIPTION:
Gestational trophoblastic disease (GTD) and gestational trophoblastic neoplasm (GTN) encompass a heterogeneous family of rare diseases that originate from fetal trophoblast cells during or after pregnancy. These diseases include benign processes with malignant potential (hydatidiform molar pregnancy) and malignancies including choriocarcinoma (CCA) and intermediate trophoblastic tumors (PSTT, ETT) . GTN more specifically includes hydatidiform molar pregnancies that have undergone malignant transformation, as well as CCA, placental site trophoblastic tumor (PSTT), and epithelioid trophoblastic tumor (ETT) . The International Federation of Gynecology and Obstetrics (FIGO) and the World Health Organization (WHO) have developed a staging and scoring system for patients with complete and partial hydatidiform molar pregnancies that have undergone malignant transformation and CCA .The scoring system is prognostic and helps guide initial treatment selection: patients with low-risk disease (i.e., a WHO score from 0 to 6) are treated with single-agent methotrexate (MTX) or dactinomycin, while patients with high-risk disease (i.e., a WHO score 7-12) are treated with multiagent regimens and ultra-high risk group; where risk score ≥12are treated with EMA-CO Despite advances in diagnosis and treatment, high-risk GTN remains a significant clinical challenge, particularly in predicting treatment response and long-term prognosis. Identifying key prognostic factors is crucial to improving therapeutic strategies and optimizing patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Patients diagnosed as high risk patient according to WHO classification[10]

  * Adequate clinical data available, including demographic, pathological, and treatment-related details.
  * Patients treated at Assuit university women's health hospital within a specified period (e.g., observational study covering period from Jan 2020 till dec 2025).

Exclusion Criteria:

* • Previous Malignancy - Patients with a history of other malignancies that may confound outcomes.

  * Non-GTN Gestational Trophoblastic Disease (GTD) - Patients with benign conditions such as complete or partial hydatidiform mole without progression to GTN.
  * Pregnant at Diagnosis - Patients diagnosed with GTN during an ongoing pregnancy.
  * Severe Comorbidities - Patients with significant non-GTN-related illnesses that could affect survival outcomes (e.g., severe heart, liver, or renal disease)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all high risk GTN patients at Assiut university women's health hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (time from treatment initiation to disease progression ,relapse ,or death from any cause) | about5-7 years from jan 2020 to dec 2027
  time from treatment initiation to disease progression ,relapse ,or death from any cause

SECONDARY OUTCOMES:
Remission cure rate | about5-7 years from jan 2020 to dec 2027
  refers to the percentage of patients who achieve complete remission, meaning the disappearance of all signs of disease, as a result of treatment. It indicates the proportion of patients who no longer show detectable evidence of the disease and remain disease-free for a specified period.
Overall survival rate. | about5-7 years from jan 2020 to dec 2027
  is the percentage of patients in a study or treatment group who are still alive after a defined period, regardless of the cause of death. It is commonly used in clinical research to measure the effectiveness of a treatment.
Recurrence (Relapse)rate | about5-7 years from jan 2020 to dec 2027
  defined as the reappearance of gestational trophoblastic neoplasia (GTN) after achieving complete remission, indicated by rising hCG levels, radiological evidence of disease, or clinical symptoms following treatment completion.
side effect of treatment protocol | about5-7 years from jan 2020 to dec 2027
Identification of number of chemotherapy courses | about5-7 years from jan 2020 to dec 2025
Identification of duration of chemotherapy courses | about5-7 years from jan 2020 to dec 2025
Identification of factors associated with poor prognosis | about5-7 years from jan 2020 to dec 2027

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Adel Aness, master degree, Principal Investigator — Assiut University; Alaa EL-Din Mahmoud Ismail, Study Director — Assiut University; Hisham Ahmed El-Sayed, Study Director — Assiut University; Mostafa Mohammed Ahmed, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyman DM, Bakios L, Gualtiere G, Carr C, Grisham RN, Makker V, Sonoda Y, Aghajanian C, Jewell EL. Placental site trophoblastic tumor: analysis of presentation, treatment, and outcome. Gynecol Oncol. 2013 Apr;129(1):58-62. doi: 10.1016/j.ygyno.2012.12.029. Epub 2012 Dec 26. PMID 23274560
- [Background] RATANAKAEW A, WASINGHON P. Prognostic Scoring and Outcome of Gestational Trophoblastic Disease Patients. J Clin Gynecol Obstet North Am. 2023 Aug;12. doi: https://doi.org/10.14740/jcgo876.
- [Background] Kong Y, Yang J, Jiang F, Zhao J, Ren T, Li J, Wang X, Feng F, Wan X, Xiang Y. Clinical characteristics and prognosis of ultra high-risk gestational trophoblastic neoplasia patients: A retrospective cohort study. Gynecol Oncol. 2017 Jul;146(1):81-86. doi: 10.1016/j.ygyno.2017.04.010. Epub 2017 Apr 29. PMID 28461032
- [Background] Liu YL, Praiss AM, Chiang S, Devereaux K, Huang J, Rizzuto G, Al-Rawi D, Weigelt B, Jewell E, Abu-Rustum NR, Aghajanian C. Gestational trophoblastic neoplasm: Patient outcomes and clinical pearls from a multidisciplinary referral center. Gynecol Oncol. 2025 Jan;192:171-177. doi: 10.1016/j.ygyno.2024.12.009. Epub 2024 Dec 13. PMID 39674133
- [Background] Lurain JR. Gestational trophoblastic disease I: epidemiology, pathology, clinical presentation and diagnosis of gestational trophoblastic disease, and management of hydatidiform mole. Am J Obstet Gynecol. 2010 Dec;203(6):531-9. doi: 10.1016/j.ajog.2010.06.073. Epub 2010 Aug 21. PMID 20728069
- [Background] El-Helw LM, Coleman RE, Everard JE, Tidy JA, Horsman JM, Elkhenini HF, Hancock BW. Impact of the revised FIGO/WHO system on the management of patients with gestational trophoblastic neoplasia. Gynecol Oncol. 2009 Jun;113(3):306-11. doi: 10.1016/j.ygyno.2009.02.006. Epub 2009 Mar 9. PMID 19269684
- [Background] Gu Y, Liu Y, Cheng H, Wang W, Xue X, Wan X, Feng F, Yang J, Ren T, Zhao J, Jiang F, Li Y, Xiang Y. Clinicopathological characteristics and oncologic outcomes of patients with gestational trophoblastic neoplasia manifesting as isolated pulmonary lesions. Gynecol Oncol. 2024 Nov;190:28-34. doi: 10.1016/j.ygyno.2024.07.686. Epub 2024 Aug 10. PMID 39128338
- [Background] Palmieri C, Dhillon T, Fisher RA, Young AM, Short D, Mitchell H, Aghajanian C, Savage PM, Newlands ES, Hancock BW, Seckl MJ. Management and outcome of healthy women with a persistently elevated beta-hCG. Gynecol Oncol. 2007 Jul;106(1):35-43. doi: 10.1016/j.ygyno.2007.01.053. Epub 2007 May 4. PMID 17482245
- [Background] Seckl MJ, Sebire NJ, Berkowitz RS. Gestational trophoblastic disease. Lancet. 2010 Aug 28;376(9742):717-29. doi: 10.1016/S0140-6736(10)60280-2. Epub 2010 Jul 29. PMID 20673583
- [Background] Ngan HY, Bender H, Benedet JL, Jones H, Montruccoli GC, Pecorelli S; FIGO Committee on Gynecologic Oncology. Gestational trophoblastic neoplasia, FIGO 2000 staging and classification. Int J Gynaecol Obstet. 2003 Oct;83 Suppl 1:175-7. doi: 10.1016/s0020-7292(03)90120-2. No abstract available. PMID 14763174
- See also: Website for a linked papers and articles — https://pubmed.ncbi.nlm.nih.gov/
- See also: Search engine that incluses files and papers similair or linked to this subject — https://scholar.google.com/
- Available data/document: papers: Not available at moment — https://pubmed.ncbi.nlm.nih.gov/ — Most of thé informations available at This site and Google Scholar